CLINICAL TRIAL: NCT03829891
Title: A Randomized, Open-label, Controlled,Parallel-group Study for Beinaglutide Versus Glargine Therapy in Glycemic Variability of Type 2 Diabetes Mellitus
Brief Title: Study for Beinaglutide Versus Glargine Therapy in Glycemic Variability of Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY20182008-1
Record Dates: First submitted 2019-01-27; First posted 2019-02-04 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2020-08

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus; Beinaglutide; glycemic variability
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — glucagon-like peptide 1 (7-36); Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beinaglutide (Experimental): 1. Beinaglutide for 8 weeks,
  2. Beinaglutide + glargine for 8 weeks(only the subjects whose blood glucose not reach the standard )
  Interventions: Drug: Beinaglutide; Drug: glargine
- glargine (Active Comparator): 1. Glargine for 8 weeks,
  2. Glargine+Beinaglutide for 8 weeks(only the subjects whose blood glucose not reach the standard )
  Interventions: Drug: Beinaglutide; Drug: glargine

INTERVENTIONS:
Drug: Beinaglutide — 1. Beinaglutide for 8 weeks,
  2. Beinaglutide + glargine for 8 weeks(only the subjects whose blood glucose not reach the standard )
Drug: glargine — 1. Glargine for 8 weeks,
  2. Glargine+Beinaglutide for 8 weeks(only the subjects whose blood glucose not reach the standard )

SUMMARY:
The investigators aimed to assess the efficacy and safety of Beinaglutide versus glargine , in individuals with type 2 diabetes who did not achieve adequate glycaemic control with oral antidiabetic drug.

DETAILED DESCRIPTION:
The investigators wonder in clinical hypoglycemic treatment for patients with hyperglycemia, whether to reduce fasting blood glucose or postprandial blood glucose first.

In this study, subjects with type 2 diabetes mellitus in combination with oral medication will be treated with basic insulin to reduce fasting blood glucose, or with beinaglutide to reduce postprandial blood glucose, in order to find out which one of controling blood glucose can be more effective and observe the change of blood fluctuation.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities
* Male or female between the age of 18 and 70 years by the time of visit 1
* Have been diagnosed as type 2 diabetes for at least half a year
* Prestudy combination OAD therapy for at least 1 month(except glinides, DPP-VI inhibitor,insulin,GLP-1 receptor agonists ),
* The dose of Sulfonylureas less than the half maximum dose of insert
* 7.5%≤HbA1c≤11.0% in recent 2 weeks or on visit 1(local lab test)
* 21Kg/m2≤BMI≤35Kg/m2

Exclusion Criteria:

* Females of child bearing potential who are pregnant, breast-feeding or intend to become pregnant or are not using adequate contraceptive methods .
* Current diagnosis or history of following:

  * Type 1 diabetes
  * Diabetes caused by impaired pancreas
  * Diabetes is the secondary diagnosis ,such as acromegaly,Cushing syndrome etc.
  * Acute decompensation of glycaemic control requiring immediate intensification of treatment to prevent acute complications of diabetes (eg. diabetes ketoacidosis, hyperosmolar coma) within 6months prior to screening.
  * Use of any glinides, DPP-VI inhibitor,GLP-1 receptor agonists within 3months prior to screening.Use of any insulin within 1months prior to screening.
  * History of allergy (such as systemic allergy, Vascular neuroedema, epidermal exfoliation, etc.)
  * Systemic use of glucocorticoids (oral or intravenous) continued for more than seven days in the past half year.
  * Triglyceride (fasting)> 4.5mmol/L at visit 1.
* Impaired liver function,such as manifested in one of the following situations:

  * Two consecutive measurements of AST or ALT in the first four weeks of the visit exceeded the maximum normal value by more than three times (local laboratory data)
  * Bilirubin synthesis and/or excretion disorders (such as hyperbilirubinemia) and other decompensated liver diseases such as coagulation,Blood disorders, hepatic encephalopathy, hypoproteinemia, ascites, esophageal variceal bleeding
  * Acute viral, active autoimmune, alcoholic and other types of hepatitis
* Moderate to severe renal impairment or end-stage renal disease (estimated kidney) at visit or 4 weeks before visit (local data)Globular filtration rate < 60 mL/minNew York Heart Association (NYHA) Class III or IV congestive heart failure
* Visit 1 has a major history of cardiovascular disease in the past three months, defined as myocardial infarction, coronary angioplasty or bypass surgery, valvular disease or repair, unstable angina, transient ischemic attack or cerebrovascular accident.
* History of acute or chronic pancreatitis
* History of gastrointestinal diseases, including gastrointestinal stoma anastomosis, intestinal resection, gastric cardiac syndrome, severe hernia, intestinal obstruction, intestinal ulcer
* Malignant tumors (except cutaneous basal cell carcinoma, cervical carcinoma in situ and prostate cancer in situ) have been diagnosed in the past five years.
* History of organ transplantation or AIDS
* History of medullary thyroid cancer
* History of alcohol or drug abuse in the past 12 months
* Individuals or researchers who do not comply with the potential risks of the program are judged to be unsuitable for the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-08-07 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-12-04 (Actual)

PRIMARY OUTCOMES:
The proportion and rate of the fasting blood glucose control. | Baseline and week 16
Proportion of patients with glycosylated hemoglobin < 7%. | Baseline and week 16
Changes of blood sugar variation . | Baseline and week 16

SECONDARY OUTCOMES:
Change percentage of glycosylated hemoglobin | Baseline and week16
Change of blood glucose | Baseline and week16
Change of blood pressure | Baseline and week16
Change of blood lipids | Baseline and week16
Change of body weight report in kilograms | Baseline and week16
Change of body mass index report in kg/m^2 | Baseline and week16
Waist-hip ration change | Baseline and week16
Oxidative Stress Indice (8-Iso-PGF2α) change | Baseline and week16
Inflammatory factors (MCP-1) change | Baseline and week16
Inflammatory factors (hs-CRP) change | Baseline and week16

OTHER OUTCOMES:
Safety Outcome Measure: Adverse Event | From baseline to week 16
  Adverse Event
Safety Outcome Measure: Serious adverse event | From baseline to week 16
  Serious adverse event

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Chang'an Hospital, Xi'an, China,Shanxi
  - Shaanxi Aerospace Hospital, Xi'an, China,Shanxi

REFERENCES:
- [Derived] Liu X, Yang W, Liu J, Huang X, Fang Y, Ming J, Lai J, Fu J, Ji Q, Wang L. The efficacy and safety of beinaglutide alone or in combination with insulin glargine in Chinese patients with type 2 diabetes mellitus who are inadequately controlled with oral antihyperglycemic therapy: A multicenter, open-label, randomized trial. J Diabetes. 2023 Oct 20;16(2):e13483. doi: 10.1111/1753-0407.13483. Online ahead of print. PMID 37864379